CLINICAL TRIAL: NCT02143869
Title: Perioperative Body Composition Changes in Patients Undergoing Gastrointestinal or Lung Cancer Surgery
Brief Title: Evolution of Corporeal Composition in the PeriOperative Period
Acronym: ECCOP
Status: Completed | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, MD, MSc, Hôpital Européen Marseille
Other Study IDs: 2013-A01346-39
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Gastrointestinal Cancer (Esophagus, Gastric, Pancreatic, Hepatic, Colorectal and Anal); Lung Cancer
Keywords: Gastrointestinal cancer; Lung cancer; Bioelectrical Impedance analysis; Body composition; Perioperative
MeSH Terms: conditions — Gastrointestinal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis — Measurements of body composition including fat mass, lean body mass, muscular mass, mineral mass, total body water, intra and extracellular water.

SUMMARY:
Denutrition and Obesity are risk factors for perioperative surgical complications.

In patient with cancer, incidence of denutrition is markedly increased. Surgical resection of cancer induces a high intensity cellular stress response and catabolism reinforcing the risk for perioperative denutrition.

In this study, we thought to investigate the change in body composition during the perioperative period using anthropometric measurements and Bioelectrical Impedance Analysis (BIA).

DETAILED DESCRIPTION:
Body composition measurements will be performed before surgical procedure (7 days) and at day 1, day 5, 1 month, 3 months and 6 months after surgery.

Others data will be recorded including anthropometric measurements, nutritional intake, occurence of surgical complication, type of surgical procedure, type and stage of cancer, and CT-scan measurements of subcutaneous abdominal fat, visceral fat and peri-renal fat before surgery and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal cancer (esophagus, gastric, pancreatic, hepatic, colorectal and anal)
* Or Lung cancer
* And planned surgical resection
* Age > 18 years

Exclusion Criteria:

* Surgical procedure planned < 48 h
* Pregnancy
* Presence of a cardiac stimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal cancer (esophagus, gastric, pancreatic, hepatic, colorectal and anal) or lung cancer undergoing curative surgical resection as part of their disease management.
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
body composition | 1 month
  The primary objective is to study the change in body composition (fat mass, lean body mass, muscular mass, mineral mass, total body water, intra and extracellular water) during the perioperative period with respect to short, mid and long term outcome.

SECONDARY OUTCOMES:
perioperative complications | 6 months
  One of the secondary objective is to investigate the relationship between baseline body composition and the occurrence of surgical complications.

OTHER OUTCOMES:
nutritional intake during perioperative period | 1 month
  One of the secondary objective is to investigate the relationship between change in body composition and perioperative nutritional intake.
cancer type and stage | 6 months
  One of the secondary objective is to investigate the relationship between baseline body composition and the type and stage of cancer.
comparison of the body composition obtained by BIA and anthropometric measurements. | 6 months
  One of the secondary objective is to compare the body composition obtained by Bioelectrical Impedance Analysis (BIA) and by anthropometric measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme ALLARDET-SERVENT, MD, MSc, Principal Investigator — Hôpital Européen Marseille
Locations (1):
- Hôpital Européen Marseille, Marseille, France